CLINICAL TRIAL: NCT05594862
Title: Treatment of Crohn's Complex Perianal Fistulas With Tissue Transplantation by Local Injection of Micro-fragmented Autologous Adipose Tissue. Multicenter Randomized Controlled Prospective Study
Brief Title: Treatment of Crohn's Complex Perianal Fistulas With Tissue Transplantation by Local Injection of Micro-fragmented Autologous Adipose Tissue.
Acronym: ATTIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lipogems International spa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATTIC
Record Dates: First submitted 2022-10-13; First posted 2022-10-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipogems (Active Comparator): surgical drainage with cone fistulectomy + infiltration of micro-fractured autologous adipose tissue at the level of the internal orifice
  Interventions: Device: Lipogems
- Placebo (No Intervention): surgical drainage with cone fistulectomy + infiltration of physiological solution and suture point positioning at the internal orifice level

INTERVENTIONS:
Device: Lipogems — Micro-fragmented adipose tissue infiltration
  Arms: Lipogems

SUMMARY:
multicentre randomized controlled prospective study aimed at evaluating the efficacy of the infiltration of microfractured adipose tissue in the healing of perianal fistulas not-responding to treatment with biologics, in order to improve the quality of life and significantly reduce the risk of definitive ostomy.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age is over 18 at the time of surgery.
* The patient suffers from Crohn's disease confirmed by instrumental and histological methods.
* The patient presents with complex perianal fistulising disease refractory to standard treatment (combination of surgical drainage of sepsis and local / systemic administration of anti-TNF-α for at least 1 year)
* The patient received, understood and signed informed consent for active participation in the study.
* The patient is able to understand the conditions of the study and to participate throughout the duration.

Exclusion Criteria:

* Patients with more than 1 internal and 3 external openings.
* Patients with ileus / colo ostomy.
* Patients with anus / rectum-vaginal fistulas.
* Patients with active HIV infections, hepatitis C (HCV), hepatitis B (HBV), tuberculosis.
* Patients with abdominal localization of Crohn's disease who may require general surgery during the study.
* Patients with active oncological or lymphoproliferative diseases from which it was not possible to safely withdraw an adequate quantity of lipoaspirate (at least 60 cc).
* Patients with clinical conditions that may compromise the success of the surgery or the follow-up.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Combined remission | 24 weeks
  The primary outcome of the study will be the evaluation of the difference between the two experimental groups in terms of "combined remission" which will be defined at 24 weeks from surgery to clinical evaluation as "absence of drainage at a slight digital compression". of all treated external orifices that were draining at baseline and pelvic MRI as the absence of abscesses> 3 mm in correspondence of the treated perianal fistulas

SECONDARY OUTCOMES:
Number of participants with Clinical remission | 2-4-8-12-24 weeks
  Comparison between the two experimental groups in terms of clinical remission at 2 weeks (± 2 days), 4 weeks (± 2 days), 8 weeks (± 2 days), 12 weeks (± 3 days) and 24 weeks ± (5 days) from surgery (ie the closure of all external orifices treated that were draining at baseline despite a slight digital compression) with the presence of abscess collections> 3 mm on MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS S Orsola Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT05594862/Prot_001.pdf